CLINICAL TRIAL: NCT03373968
Title: Open Label, Long-term Safety, Tolerability, and Efficacy Study of GIVINOSTAT in All DMD Patients Who Have Been Previously Treated in One of the GIVINOSTAT Studies
Brief Title: Givinostat in Duchenne's Muscular Dystrophy Long-term Safety and Tolerability Study
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Collaborators: Cromsource (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSC/14/2357/51
Record Dates: First submitted 2017-12-04; First posted 2017-12-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — givinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- givinostat (Experimental): Givinostat oral suspension (10 mg/mL) twice daily in a fed state
  Interventions: Drug: Givinostat

INTERVENTIONS:
Drug: Givinostat — suspension of givinostat (10 mg/mL)

SUMMARY:
This is an open label, long-term safety, tolerability, and efficacy study of GIVINOSTAT in all DMD (Duchenne's muscular dystrophy) patients who have been previously treated in one of the GIVINOSTAT studies.

DETAILED DESCRIPTION:
GIVINOSTAT oral suspension (10 mg/mL) has to be administered orally as 2 oral doses daily while the subject is in a fed state. The starting dose of GIVINOSTAT in the present long term study will be the same that the subject was receiving at the end of the previous DMD GIVINOSTAT study.

As weight affects GIVINOSTAT exposures, the dosage will be modified based on subject weight according the rules detailed in the study protocol section 11.2.2.1.

In addition, in case a subject will have a consistent (e.g., at least 2 consecutive evaluations) platelets count ≤150 x 10^9/L and not meet the stopping criteria for platelets, the Investigator will have to reduce the dose of 1/3 or 20% less of the current dose as described in the study protocol section 10.5.1.3. During the first month of treatment, platelets count assessment will be performed weekly, while during the second month it will be performed every 2 weeks, in order to strictly monitor this parameter for safety reasons, with the exclusion of subjects coming from study DSC/11/2357/43 for which the first visit will be 4 months after the Visit 1/baseline visit.

Study drug should be permanently interrupted if any of the following occurs:

* severe drug-related diarrhoea (i.e., increase of ≥7 stools per day);
* any drug-related SAE;
* QTcF >500 msec;
* platelets count ≤50 x 10^9/L;
* white blood cells ≤2.0 x 10^9/L;
* hemoglobin ≤8.0 g/dL; To avoid laboratory errors and anomalous values, test must be confirmed with a repeated test performed on the next working day. The treatment should be stopped until the retest result becomes available. If the repeated test is still under the stopping limit value, study drug must be permanently discontinued. If the repeated test is acceptable, the subject can resume treatment.

The Investigator will follow up the patient until resolution or acceptable stabilization of the event occurs and document all the relevant information, as applicable. After the resolution/stabilization of the event, the subject will be withdrawn from the study and the EOS Visit (see Section 12.1.10) will be performed.

Any decision relevant to the dose adjustment and/or modification of schedule of assessments can be discussed with the Medical Monitor, but the final decision remains with the Investigator only or its authorized designee.

ELIGIBILITY:
Inclusion Criteria:

1. Must have participated in one of the previous studies with GIVINOSTAT in DMD and have attended the End of Study Visit or must have been screened in study DSC/14/2357/48 and met:

   * all the inclusion criteria and none of the exclusion criteria,
   * had a baseline vastus lateralis muscle fat fraction (VL MFF) assessed by MRS in the range ≤5% or >30%, i.e. included in"off-target" group,
   * never been randomized because, the enrollment in the off target group was completed.
2. Aged ≥6 years old;
3. Are able to give informed assent and/or consent in writing signed by the subject and/or parent/legal guardian (according to localregulations);
4. Subjects must be willing to use adequate contraception:

   * Contraceptive methods must since the previous GIVINOSTAT study through 3 months after the last dose of study drug, and include the following:

     * True abstinence (absence of any sexual intercourse), when in line with the preferred and usual lifestyle of the subject.
     * Periodic abstinence (e.g. calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception.
     * Condom with spermicide and the female partner must use an acceptable method of contraception, such as an oral,
     * transdermal, injectable or implanted steroid-basedcontraceptive, or a diaphragm or a barrier method of contraception in conjunction with spermicidal jelly such asfor example cervical cap with spermicide jelly.

Exclusion Criteria:

1. Use of any pharmacologic treatment, other than corticosteroids, that might have had an effect on muscle strength or function within 3 months prior to be enrolled in this study (e.g., growth hormone); Vitamin D, calcium, and any other supplements will be allowed;
2. Use of any current investigational drug other than Givinostat;
3. Have presence of other clinically significant disease, which, in the Investigator's opinion, could adversely affect the safety of the subject, making it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results;
4. Have a diagnosis of other uncontrolled neurological diseases or presence of relevant uncontrolled somatic disorders that are not related to DMD;
5. Have platelets count, White Blood Cell and Hemoglobin at screening < Lower Limit of Normal (LLN)* (for abnormal screening laboratory test results (<LLN), the platelets count, White Blood Cell and Hemoglobin will be repeated once; if the repeat test result is still <LLN, then exclusionary);
6. Have Triglycerides > 300 mg/dL (3.42 mmol/L) in fasting condition at screening visit* (for abnormal screening laboratory test results (>300 mg/dL), the triglycerides will be repeated once; if the repeat test result is still >300 mg/dL, then exclusionary);
7. Have inadequate renal function, as defined by serum Cystatin C >2 x the upper limit of normal (ULN) at screening visit*. If the value is >2 x ULN, the serum Cystatin C will be repeated once; if the repeated test result is still >2 x ULN, the subject should be excluded);
8. Have heart failure (New York Heart Association Class III or IV)
9. Have a current liver disease or impairment, including but not limited to an elevated total bilirubin* (i.e. > 1.5 x ULN), unless secondary to Gilbert disease or pattern consistent with Gilbert's;
10. Have a baseline QTcF >450 msec, (as the mean of 3 consecutive readings 5 minutes apart) or history of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, or family history of long QT syndrome);
11. Have a psychiatric illness/social situation rendering the potential subject unable to understand and comply with the muscle function tests and/or with the study protocol procedures.
12. Have any hypersensitivity to the components of study medication;
13. Have a sorbitol intolerance or sorbitol malabsorption or have the hereditary form of fructose intolerance.

    * the Investigators to evaluate these exclusion criteria can use the laboratory results obtained within 5 months from V1, to allow the continuity of the treatment. It is worth noting, as soon as the site will receive the laboratory results done in screening/baseline (Visit 1) visit they will check the GIVINOSTAT dose and modify it as per protocol safety rules and/or dosage modifications rules.

Min Age: 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2017-10-24 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Through study completion, an average of 1 year
  Type, incidence, and severity of treatment related/not related adverse events(AEs) and serious adverse event (SAEs)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (10):
  - University of California - Davis Medical Center - Devis Physical Medicine & Rehabilitation, Sacramento, California
  - Rady Children's Hospital center - UCSD Department of Neuroscience, San Diego, California
  - Connecticut Children's Medical Center, Neurology Division, Hartford, Connecticut
  - Child Health Research Institute, Gainesville, Florida
  - MD Rare Disease Research, LLC, Atlanta, Georgia
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Washington University School of Medicine in St Louis Department of Neurology 660 S.Euclid Avenue, Campus Box 8111, St Louis, Missouri
  - Shriners Hospitals for Children, Portland, Oregon
  - The Children's Hospital of Philadelphia Colket Translational Research Building, Philadelphia, Pennsylvania
  - Virginia Commonwealth University Childrens Hospital of Richmond at, Richmond, Virginia
- Belgium (2):
  - University Hospitals Leuven, Neuromuscular Reference Centre, Child Neurology, Leuven
  - Hospital de La Citadelle, Centre de Référence des Maladies Neuromuscolaires (CRMN), Liège
- Canada (3):
  - Kinsmen Research Centre - Alberta Children's Hospital, Calgary, Alberta
  - The University of British Columbia, Children's and Womens Health Centre of BC Branch, Vancouver, British Columbia
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario
- France (2):
  - CHU de Nantes - Hotel-Dieu - Hopital Nord Laennec, rez-de-chausse haut ail Ouest, Nantes
  - Hôpital Armand Trousseau I-Motion - Plateforme d'essais cliniques pédiatriques Bâtiment Lemariey - Porte 20 * 2ème étage 26 Avenue du Dr Arnold Nette, Paris
- Germany (3):
  - Universitätsklinikum Essen - Kinder-und Jugendmedizin Neuropadiatrie, Essen
  - Klinik- und Poliklinik fur Kinder- und Jugendmedizin, Universitatsklinikum HamburgEppendorf, Martinistr. 52, Hamburg
  - Klinikum der Universitat Munchen, Campus Innenstadt, Lindwurmstr. 4, München
- Institute of Neurology - Schneider Children's Medical Center of Israel Kaplan, 14, Petah Tikva, Israel
- Italy (7):
  - U.O.S.D. Centro Traslazionale di Miologia e Patologie Neurodegenerative, Building 16 - ground floor IRCCS Istituto Giannina Gaslini,, Genova
  - A.O.U. Policlinico G. Martino, U.O.C. Neurologia e Malattie Neuromuscolari, Messina
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, UOS di Neurologia Pediatrica, Milan
  - IRCCS Istituto Neurologico Carlo Besta, Milan
  - Centro Clinico NeMO Fondazione Serena ONLUS Area SUD, Milan
  - Ospedale Pediatrico Bambino Gesù, Malattie Neuromuscolari e Neurodegenerative, Roma
  - Fondazione Policlinico Universitario "A.Gemelli", UOC Neuropsichiatria Infantile, Roma
- Netherlands (2):
  - Leiden University Medical Center LUMC, Albinusdreef 2, Leiden
  - Radboud University Medical Centre, Nijmegen
- Clinic of Neurology and Psychiatry for Children and Youth - Neurology Department Dr. Subotic 6a,, Belgrade, Serbia
- Spain (4):
  - Neuromuscular Pathology Unit - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcellona
  - Hospital Materno-Infantil, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politècnic La Fe - Servicio Neurologia, Valencia
- United Kingdom (4):
  - Alder Hey Children's Hospital NHS Trust, Liverpool, UK
  - The Robert Jones and Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Gobowen
  - UCL Great Ormond Street Institute of Child Health, Dubowitz Neuromuscular Centre and MRC Centre for NMD, London
  - The John Walton Muscular Dystrophy Research Centre, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McDonald CM, Guglieri M, Vucinic D, Acsadi G, Brandsema JF, Bruno C, Finanger EL, Harper A, Lobato ML, Masson R, Muelas N, Munell F, Nevo Y, Pereon Y, Phan H, Sansone VA, Scoto M, Willis T, Finkel RS, Vandenborne K, Cazzaniga S, Montrasio S, Alessi F, Bettica P, Mercuri E; Givinostat Study 51 Investigators; Cooperative International Neuromuscular Research Group (CINRG) Duchenne Natural History Study (DNHS) Investigators; ImagingDMD Investigators. Long-Term Evaluation of Givinostat in Duchenne Muscular Dystrophy, and Natural History Comparisons. Ann Clin Transl Neurol. 2025 Nov;12(11):2335-2348. doi: 10.1002/acn3.70165. Epub 2025 Aug 19. PMID 40830818